CLINICAL TRIAL: NCT01174836
Title: Patient and Physician Attitudes About Informed Consent for Emergency Department (ED) Computerized Axial Tomography (CT) Scans
Acronym: CT Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-0807
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Attitudes About CT Utilization
Keywords: CT utilization; physician attitudes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Educational session — Physicians will have a brief education session provided in powerpoint about the risks of CT

SUMMARY:
Hypothesis: The majority of Emergency physicians and patients do not feel that specific informed consent should be obtained for ED CT scans.

Secondary Hypothesis: Emergency attending physicians and residents will have similar attitudes about CT scan consent issues. Physician attitudes toward obtaining consent for CT scans will change after an educational program about the associated risks.

DETAILED DESCRIPTION:
ED residents and ED attendings who attend grand rounds will be given a survey and asked to anonymously complete the first portion before grand rounds (Figure 1, example A). The first portion will assess basic demographics, CT ordering patterns and experiences, and attitudes about informed consent. They will be provided with an educational program at grand rounds that reviews current literature relevant to CT utilization and consent issues. After the lecture they will be asked to complete the second section of the survey (Figure 1, Example B). Both portions of the survey will be simultaneously returned in a sealed envelope and placed in a collection box at grand rounds.

ED attendings who do not attend grand rounds will only be asked to complete the first portion of the survey (Figure 1, example A). Resident or attending consent to participate will not be coerced, and participation will be implied by completion of the survey.

ELIGIBILITY:
Inclusion Criteria:

* Current ED resident and attending physicians
* An ED patient (or their surrogate) that is able to understand and respond in writing to the questions given.

Exclusion Criteria:

* Anyone who declines to participate.
* An ED patient who is not able to understand questions or respond in writing to the questions given (and does not have a surrogate that understands questions and respond in writing to the questions given).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Survey response to physician attitudes about ordering CT | 30 minutes (after lecture) resurvey
  Before and after education physicians will be surveyed as to the attitudes about ordering ct's